CLINICAL TRIAL: NCT01769781
Title: Treatment of Patients With Endometriosis Recurrence With Aromatase Inhibitor (Anastrazole) Plus GnRH-agonist (Luprolide).
Brief Title: Anastrazole Plus GnRH-agonist in the Treatment of Endometriosis Recurrence
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Centre for Endocrinology and Reproductive Medicine, Italy (Network)
Responsible Party: Principal Investigator, Fabio Scarpellini, PRINCIPAL INVESTIGATOR, Centre for Endocrinology and Reproductive Medicine, Italy
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CR013-01
Record Dates: First submitted 2013-01-15; First posted 2013-01-17 (Estimated); Last update posted 2016-04-27 (Estimated); Status verified 2016-04

CONDITIONS: Endometriosis
Keywords: endometriosis recurrence; pelvic pain; aromatase inhibitor
MeSH Terms: conditions — Endometriosis; Pelvic Pain | interventions — Anastrozole; Gonadotropin-Releasing Hormone

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- anastrazole (Experimental): women with endometriosis recurrence will be treated with Leuprolide acetate 11,25mg plus anastrazole 1mg/day for three months
  Interventions: Drug: anastrazole
- GnRH analog alone (Active Comparator): women with endometriosis recurrence will be treated with leuprolide acetate 11.25mg
  Interventions: Drug: GnRH analog alone

INTERVENTIONS:
Drug: anastrazole — combined treatment with aromatase inhibitor (anastrazole) plus GnRH analog (leuprolide acetate) for three months
  Arms: anastrazole
Drug: GnRH analog alone — treatment for three months with GnRH analog (leuprolide acetate) alone
  Arms: GnRH analog alone

SUMMARY:
The aromatase inhibitor (anastrazole) plus long acting GnRH agonist leuprolide acetate will be tested for the treatment of women with endometriosis recurrence compared with classical GnRH analog treatment. Pain symptom disappearance and disease free time during follow-up will be the outcomes for establishing which medical treatment is the best in endometriosis recurrence treatment.

DETAILED DESCRIPTION:
Endometriosis is a chronic disease affecting 5-10% of women in reproductive age, showing recurrence after surgery at least in 20-50% after 5 years of follow-up. Aromatase inhibitor plus GnRH analog may be more effective than GnRH agonist alone in the treatment of endometriosis recurrence.

ELIGIBILITY:
Inclusion Criteria:

* women affected by endometriosis showing recurrence of pain symptoms, previous surgery for endometriosis

Exclusion Criteria:

* presence of other systemic diseases

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 70 (Actual)
Dates: Start 2013-01; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
disease free time | 24 months
  time without pain symptoms due to the disease recurrence

SECONDARY OUTCOMES:
time of pain disappearance | 24 months
  time needed during treatment to improve pain symptoms

OTHER OUTCOMES:
reduction of endometriosis lesions | 24 months
  endometriosis lesions regression during treatment evidenced by MRI scan

CONTACTS AND LOCATIONS:
Overall Officials: marco sbracia, md, Study Chair — CERM-HUNGARIA
Locations (1):
- Cerm-Hungaria, Rome, Italy